CLINICAL TRIAL: NCT02948257
Title: Multi-center, Prospective, PM Registry for Procedural Outcomes Using the Cardiva VASCADE VCS for Closing the Femoral Arteriotomy After Percutaneous Endovascular Procedures Via Antegrade Access.
Brief Title: VASCADE ANTEGRADE-PVD Post-Market Registry
Status: Completed | Type: Observational
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL 0502-02
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Surgical Wound
Keywords: Vessel closure; Antegrade access; Femoral arteriotomy; Peripheral endovascular interventions
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiva Medical VASCADE VCS — At the end of peripheral endovascular interventional procedures performed via an antegrade femoral arterial approach, the femoral arterial access site is closed with the VASCADE VCS to achieve arterial hemostasis.

SUMMARY:
The objective of the registry is to collect procedural outcomes data when the Cardiva VASCADE Vascular Closure System (VCS) is used to seal femoral arterial access sites at the completion of ipsilateral peripheral interventional procedures performed through 5-7F introducer sheaths via an antegrade approach.

DETAILED DESCRIPTION:
Due to the growing adoption of antegrade femoral access and the use of VCDs to close these arteriotomies, it is important to collect performance and complication outcomes data related to this procedural variable. The aim of this registry is to consistently collect prospective data on procedural outcomes on antegrade access cases closed with the VASCADE VCS in a way that is consistent with the RESPECT Study design and the FDA-approved Instructions for Use (IFU).

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for post-procedural manual compression
* Able to ambulate at least 20 feet, with or without assistance

Exclusion Criteria:

* Active systemic or cutaneous infection or inflammation
* Ipsilateral femoral arteriotomy with any of the following conditions: a) access within < or = 10 days; b) any residual hematoma, significant bruising, or known associated vascular complications; or c) within < or = 90 days, use of an intra-vascular closure device (i.e., Angioseal)
* Previous vascular grafts or surgery at the target vessel access site
* Major amputation of ipsilateral lower extremity - previous history of, or planned within next 30 days prior to study exit
* Extreme morbid obesity (BMI greater than 4 kg/m2) or underweight (BMI less than 20 kg/m2)
* Femoral arterial diameter < 6 mm at access site
* Antegrade arterial access site is a side stick and/or is not a single anterior wall femoral puncture
* Length of tissue tract, the distance between the anterior arterial wall and skin, is < 2.5 cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acceptable candidate for an elective, non-emergent ipsilateral peripheral interventional endovascular procedure via antegrade access of the femoral artery using a 5, 6 or 7 Fr introducer sheath
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Shishehbor, MD, Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (5):
  - Cardiovascular Institute of the South, Houma, Louisiana
  - North MS Medical Center, Tupelo, Mississippi
  - Coastal Surgery Specialists, Wilmington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - San Antonio Endovascular and Heart Institute, San Antonio, Texas

REFERENCES:
- [Background] Hermiller JB, Leimbach W, Gammon R, Karas SP, Whitbourn RJ, Wong SC, Goswami N, McCabe J, Cavros NG, Paulus R, Naidu SS, Turi ZG. A prospective, randomized, pivotal trial of a novel extravascular collagen-based closure device compared to manual compression in diagnostic and interventional patients. J Invasive Cardiol. 2015 Mar;27(3):129-36. PMID 25740963

RESULTS

PARTICIPANT FLOW:
Groups:
- VASCADE VCS: The Cardiva VASCADETM Vascular Closure System (VCS) was used to seal femoral arterial access sites at the completion of ipsilateral peripheral interventional procedures performed through 5-7 Fr introducer sheaths via an antegrade approach.
Period: Overall Study
Arm/Group | VASCADE VCS
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (4.46)

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis (TTH)
Description: Time to Hemostasis (TTH) is defined as elapsed time between VASCADE device removal and first observed and confirmed arterial hemostasis.
Time Frame: Procedural, usually within 15 minutes of enrollment
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
minutes | 5.87 (2.44)

2. Primary Outcome: Major Access Site Closure-related Complications
Description: Patient incident rate of combined major access site closure-related complications through 30 days
Time Frame: Through 30 days +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
Participants | 1

3. Secondary Outcome: Time to Ambulation (TTA)
Description: Time to Ambulation (TTA) is defined as elapsed time between VASCADE device removal and when subject stands and walks 20 feet without evidence of arterial re-bleeding from the access site.
Time Frame: Prior to discharge, usually within 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
hours | 4.48 (3.83)

4. Secondary Outcome: Time to Discharge (TTD)
Description: Time to Discharge (TTD) is defined as elapsed time between VASCADE device removal and discharge from the facility.
Time Frame: Through hospital discharge, usually within 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
hours | 5.97 (5.85)

5. Secondary Outcome: Device Success
Description: Device Success is defined as the ability to deploy the delivery system, deliver the collagen, and achieve hemostasis with the Cardiva VASCADE VCS alone or with adjunctive compression.
Time Frame: Procedural, usually within 15 minutes of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
Participants | 51

6. Secondary Outcome: Procedure Success
Description: Procedure Success is defined as attainment of Device Success and freedom from major access site closure-related complications through 30 days.
Time Frame: Through 30 +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 51
Participants | 50

7. Secondary Outcome: Minor Access Site Closure-related Complications
Description: Patient incident rate of combined minor access site closure-related complications through 30 days
Time Frame: Through 30 +/- 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | VASCADE VCS
Number analyzed (Participants) | 52
Participants | 51

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | VASCADE VCS
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 2/52
Other Adverse Events (participants affected / at risk) | 11/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VASCADE VCS (N=52)
Chronic osteomyelitis of ankle/foot (Infections and infestations) | 1 (1) — Chronic osteomyelitis of ankle/foot
Anemia (Blood and lymphatic system disorders) | 2 (2) — Anemia
Sepsis (Infections and infestations) | 1 (1) — Sepsis
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Acute Kidney Injury
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VASCADE VCS (N=52)
Access site arterial re-bleeding after initial hemostasis (Blood and lymphatic system disorders) | 1 (1) — Access site arterial re-bleeding after initial hemostasis
Residual hematoma < 6 cm (Blood and lymphatic system disorders) | 2 (2) — Residual hematoma < 6 cm
Tissue tract oozing - prolonged (Infections and infestations) | 2 (2) — Tissue tract oozing - prolonged
Pseudoaneurysm not requiring repair (Cardiac disorders) | 1 (1) — Pseudoaneurysm not requiring repair
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) — Bruising
Groin pain (Surgical and medical procedures) | 1 (1) — Groin pain
Angina (Cardiac disorders) | 1 (1) — Angina
Worsening PVD (Vascular disorders) | 4 (4) — Worsening PVD
Hypotension (Cardiac disorders) | 1 (1) — Hypotension
Mechanical Fall (General disorders) | 1 (1) — Mechanicall Fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02948257/Prot_SAP_ICF_000.pdf